CLINICAL TRIAL: NCT03999164
Title: Imaging of Glial Activation and Risk for Post-Traumatic Epilepsy
Brief Title: Imaging of Neuro-Inflammation and the Risk for Post-Traumatic Epilepsy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1437948
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Epilepsy, Post-Traumatic
Keywords: neuroinflammation; activated microglia; TSPO; Traumatic Brain Injury; TBI; Positron emission tomography
MeSH Terms: conditions — Epilepsy, Post-Traumatic; Neuroinflammatory Diseases; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Moderate to Severe Traumatic Brain Injury (Experimental): All patients will undergo a [18F]DPA-714 PET scan of the brain 2 weeks and 2 months following moderate to severe traumatic brain injury to quantify neuroinflammation.
  Interventions: Drug: [18F]DPA-714 Positron Emission Tomography Scan

INTERVENTIONS:
Drug: [18F]DPA-714 Positron Emission Tomography Scan — All patients will undergo a [18F]DPA-714 PET scan of the brain 2 weeks and 2 months following moderate to severe traumatic brain injury to quantify neuroinflammation.

SUMMARY:
This study plans to evaluate the time course of inflammation in the brain after a moderate to severe traumatic brain injury using positron emission tomography (PET) brain imaging. Patients will undergo PET scans of the brain at two weeks and two months after injury to measure neuro-inflammation. The results of the PET scans will be analyzed and correlated with the risk of post-traumatic epilepsy.

DETAILED DESCRIPTION:
The development of post-traumatic epilepsy (PTE) is associated with neurobiological, cognitive, psychological, and social consequences that are far-reaching for the patient. Despite our keen awareness of this significant public health issue, little is known regarding the biological mechanisms leading to PTE. One plausible mechanism is that unchecked neuroinflammation, a process that occurs in animal and human models of both traumatic brain injury (TBI) and epilepsy, leads to altered synaptic transmission and neuronal excitability. However, the direct relationship between neuroinflammation and PTE has been difficult to ascertain from pre-clinical studies as they may not accurately reflect the human condition, as few animal models can induce the progression of PTE without a pharmacological enhancer and are predominately limited to studies of mild-to-moderate TBI given high animal mortality rates from more severe injuries. Measurements of neuroinflammation in human TBI and epilepsy has also proven difficult without invasive monitoring or post-mortem evaluations, and measurements of inflammatory mediators in blood or serum may not meaningfully reflect the extent of neuroinflammation.

Encouragingly though, positron emission tomography (PET) can be used to measure the degree of in vivo glial activation in the central nervous system through radiotracer binding of the translocator protein (TSPO), serving as a surrogate of neuroinflammation. Minimally expressed in the uninjured brain, TSPO binding is increased in a number of brain disorders associated with neuroinflammation, including Alzheimer's disease, ischemic stroke, recurrent head trauma in football, brain metastases, TBI, and epilepsy, and is expressed predominately by activated microglia, the main mediators of neuroinflammation. Currently, no pre-clinical or clinical study has analyzed the relationship between glia activation, as measured by TSPO PET, and the risk for developing PTE. Accordingly, we plan to use [18F]DPA-714 to characterize neuro-inflammation following moderate-to-severe TBI in order to better understand the temporal time course of neuro-inflammation following injury and its potential role in epileptogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Acute Traumatic Brain Injury (TBI)
* Age 18-100 are eligible
* Glasgow Coma Scale (GCS) 3-13 without continuous sedation at time of enrollment
* Ability to enroll within 72 hours of injury
* Hemorrhagic contusional injuries to frontal and/or temporal lobes.
* Polytrauma including long bone fractures, blunt trauma, abdominal trauma or similar will be allowed
* Penetrating TBI if continuous electroencephalography (cEEG) is feasible and survival for 2 years is feasible, recognizing that MRI may not be feasible with some forms of penetrating trauma

Exclusion Criteria:

* Low-affinity TSPO binding profile
* Ages 17 years or younger
* Patients with diffuse axonal injury in the absence of hemorrhagic contusions or skull fracture, and isolated epidural hemorrhages that improve after evacuation
* No planned continuous EEG monitoring during injury day 1-7
* Inability to undergo MRI at 14 days (± 4 days) due to bullet, metal implant, or pacemaker
* Pregnancy
* Pre-existing Neurodegenerative Disorders
* Pre-existing epilepsy/seizure disorder
* Pre-existing dementia
* Isolated anoxic brain injury
* Incarceration present or pending
* Devastating cervical spine injury

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2026-08-14 (Estimated); Study Completion 2026-08-14 (Estimated)

PRIMARY OUTCOMES:
Quantification of [18F]DPA-714 binding in the brain following moderate to severe traumatic brain injury | 2 weeks
Quantification of [18F]DPA-714 binding in the brain following moderate to severe traumatic brain injury | 2 months

SECONDARY OUTCOMES:
Frequency of early seizures, epileptiform discharges, and post-traumatic epilepsy | Admission - two years
Modified Rankin Scale | 3 and 6 months
  All patients will undergo a phone survey at 3 and 6 months post-injury to assess functional outcome using the Modified Rankin Scale. The Modified Rankin Scale measures the degree of disability or dependence in daily activities of patients who have suffered an neurological injury, ranging from 0 (no symptoms) to 6 (dead).
Quantify the association between contusion volume and adjacent cerebral edema with [18F]DPA-714 binding on PET scans | 2 weeks
  All patients will undergo multi-modal MRI brain (Fluid-attenuated inversion recovery (FLAIR), susceptibility weighted imaging(SWI), diffusion weighted imaging(DWI)) two weeks post-injury to assess for acute structural abnormalities

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No